CLINICAL TRIAL: NCT06051162
Title: Effect of Use of Hypotension Prediction System in Prevention of Postoperative Acute Kidney Injury in Robotic-assisted Urologic Surgery
Brief Title: HPI Effect in Robotic Urological Surgery on AKI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ewha Womans University Mokdong Hospital (Other)
Responsible Party: Principal Investigator, Sooyoung Cho, Assistant Professor, Ewha Womans University Mokdong Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-02-016-003
Record Dates: First submitted 2023-09-17; First posted 2023-09-22 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer; Renal Cancer; Urologic Diseases
Keywords: Robotic
MeSH Terms: conditions — Prostatic Neoplasms; Kidney Neoplasms; Urologic Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPI (Experimental): Managing intraoperative hemodynamic condition under the HPI guidance
  Interventions: Device: BP management with HPI guidance
- Control (No Intervention): Managing intraoperative hemodynamic condition with standard anesthesia care (blinding the HPI monitor screen)

INTERVENTIONS:
Device: BP management with HPI guidance — The hemodynamic condition of the HPI group will be managed by HPI guidance which is derived by arterial pressure waveform information, including Eadyn, SVV, dP/dt.
  Arms: HPI

SUMMARY:
It is a single-center randomized controlled trial that aims to figure out the effect of the hypotension prediction index (HPI) on the prevention of acute kidney injury (AKI) after robot-assisted urological surgery. The primary hypothesis is that HPI software guidance prevents postoperative AKI by reducing the duration and severity of intraoperative hypotension (IOH).

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 19
* Patients undergoing robot-assisted urological surgery

Exclusion Criteria:

* Unable to voluntarily give consent
* Unable to use both radial arteries due to such reasons: prior surgery on the radial artery, breast cancer history with axillary LN dissection, AV fistula for renal replacement therapy, or abnormal Allen's test.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury | Seven day after the operation
  Occurrence of acute kidney injury after robotic urological surgery

SECONDARY OUTCOMES:
Depth and duration of hypotension | From applying HPI (hypotension prediction index) monitor to the arterial line to the end of the anesthesia
  Depth and duration of hypotension will be assessed by calculating time weighted average (TWA) of hypotension under mean arterial pressure under 65 mmHg during the operation
Hypotension prediction index | From applying HPI (hypotension prediction index) monitor to the arterial line to the end of the anesthesia
  Time weighted average of hypotension prediction index during the operation
Biomarkers | Baseline, immediate postop
  Biomarkers for early detection of AKI - Cystacin C, KIM-1

CONTACTS AND LOCATIONS:
Locations (1):
- Ewha Womans University Mokdong Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No